CLINICAL TRIAL: NCT01489722
Title: A Phase Ia/Ib, Open-Label, Multicentre, Two-Part Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of AZD1208 Administered Daily in Adult Patients With Recurrent or Refractory Acute Myelogenous Leukemia (AML)
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of AZD1208 in Acute Myelogenous Leukemia (AML) Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4510C00001
Record Dates: First submitted 2011-11-22; First posted 2011-12-12 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; AML; AZD1208
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — AZD1208

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD1208 (Experimental): Single ascending dose escalation of 3 - 6 patient cohorts until maximum tolerated dose (MTD) is established. Up to 12 patients may be included at any dose not determined to be intolerable. Safety expansion using MTD in up to 44 Acute myelogenous leukemia (AML) patients.
  Interventions: Drug: AZD1208

INTERVENTIONS:
Drug: AZD1208 — Daily oral doses of AZD1208 for 28 day cycles until progression or unacceptable toxicity develops. Starting dose will be 120 mg and will be escalated in successive cohorts until an MTD is established.

SUMMARY:
The purpose of this open label study is to evaluate the safety, tolerability, pharmacokinetics, and efficacy of AZD1208 in patients with recurrent or refractory Acute Myelogenous Leukemia (AML). This study will have two parts. In Part A, patients will receive escalating doses to identify the maximum tolerated dose (MTD). In Part B, the efficacy of the maximum tolerated dose will be evaluated in a expanded group of patients.

DETAILED DESCRIPTION:
A Phase Ia/Ib, Open-Label, Multicentre, Two-Part Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of AZD1208 Administered Daily in Adult Patients with Recurrent or Refractory Acute Myelogenous Leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age
* Patients with relapsed or refractory Acute myelogenous leukemia (AML) or AML secondary to myelodysplastic syndromes, myeloproliferative neoplasm, or chronic myelogenous leukemia
* Eastern Oncology Cooperative Group (ECOG) performance status 0-2 and considered likely to complete at least 4 weeks of therapy

Exclusion Criteria:

* With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment.
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and HIV.
* Active heart disease including myocardial infarction within the last 3 months, symptomatic coronary artery disease, clinically significant arrhythmias not controlled by medication or uncontrolled congestive heart failure
* Prior allogeneic transplant requiring immunosuppressive therapy (Patients with prior allogeneic transplants who remain clinically stable for ≥ 2 weeks or more off immunosuppressive therapy, are eligible)
* White blood cell count ≥ 100,000/mm3 (100x10*9/L)
* Type 1 Diabetes or uncontrolled Type II Diabetes
* HbA1C ≥8% or fasting blood glucose >160 mg/Dl (>8.9 mmol/L)
* Baseline fasting total cholesterol >300 mg/dL (>7.75 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Part A: Number of patients with dose limiting toxicities (DLTs) [Maximum Tolerated Dose (MTD) is defined as the maximum dose level below the dose level at which ≥ 33 % of at least 6 patients of a cohort experience DLTs during cycle 1.] | 28 days (cycle 1)
Part B: Number of patients with Complete Remission (CR) or CR with incomplete blood count recovery (CRi) | From baseline until disease progression or discontinuation from study (expected duration of treatment: approximately 3 months)

SECONDARY OUTCOMES:
Part A and B: Number of patients with adverse events and serious adverse events | From cycle 1 day 1 until treatment discontinuation (expected duration of treatment: approximately 3 months)
Part A and B: Description of the pharmacokinetics (PK) of AZD1208 in terms of area under plasma concentration-time curve(AUC), maximum plasma concentration (Cmax), and time to maximum plasma concentration (Tmax) | Cycle 1Day 1- pre-dose through 24 hours post dose and Cycle 1 Day 14 - pre-dose through 24 hours post-dose. Interval timepoints : predose, 30 mins, 1 hour(hr), 1.5hr, 2hr , 3hr, 6hr , 8hr, 24 hours and at same timepoints at Cycle 1 Day 14.
Part A and B: Description of urine pharmacokinetics (PK) of AZD1208 in terms of the cumulative amount of drug excreted unchanged into urine from zero to time and renal clearance | Cycle 1Day 1- pre-dose through 24 hours post dose and Cycle 1 Day 14 - pre-dose through 24 hours post-dose.during 0 - 24 hours after dosing.
Part A and B: Number of patients with response of Complete Remission(CR), CR with incomplete blood count recovery, Partial Remission, or Morphologic Leukemia-Free | From baseline until disease progression or discontinuation from study (expected duration of treatment: approximately 3 months)
Part B: Duration of CR or CRi based on time from first documentation of CR to relapse | From baseline until disease progression or discontinuation from study (expected duration of treatment: approximately 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Neumann, MD, Study Director — Sponsor GmbH
Locations (4):
- United States (3):
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Houston, Texas
- Research Site, Toronto, Ontario, Canada

REFERENCES:
- See also: D4510C00001_CSR_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1500&filename=D4510C00001_CSR_Synopsis.pdf